CLINICAL TRIAL: NCT00067678
Title: Soy Protein in Early Diabetic Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000323-01 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Diabetic Nephropathy; Diabetes Mellitus
Keywords: diabetic nephropathy; nephropathy; diabetes; diabetes mellitus; type I diabetes; soy protein
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases; Diabetes Mellitus, Type 1 | interventions — Soybean Proteins

INTERVENTIONS:
Drug: soy protein

SUMMARY:
Diabetic nephropathy is a frequent cause of end-stage renal disease. Reduction of dietary protein has been used to slow down renal disease progression, but patients are often unwilling to make these dietary changes. Other research suggests that changing the quality of dietary protein may be as effective as reducing the total amount of ingested protein. This study hopes to show that soy protein, a plant protein relatively high in essential amino acids and with high nutritional value, maye be beneficial to Type I diabetic patients with incipient renal disease.

ELIGIBILITY:
Inclusion criteria:

* Age 18-40;
* Diabetic nephropathy;
* Type I diabetes mellitus.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2001-07; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fanti, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States